CLINICAL TRIAL: NCT02915497
Title: A Pilot Randomized Controlled Trial in Patients Within One Week of Acute Physical Trauma to Test the Feasibility and Effectiveness of AEPET Plus RBT Versus RBT Alone for the Prevention of PTSD and Depression
Brief Title: Early Prevention of PTSD in Patients Within One Week of Acute Physical Trauma
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary data analysis underway, will determine whether additional recruitment is necessary upon review of collected data.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 411-2014
Record Dates: First submitted 2016-07-14; First posted 2016-09-27 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Prolonged Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment As Usual + Resilience-Based Supportive Therapy (No Intervention): Routine psychosocial management of trauma patients, including Manualized Resilience-Based Therapy.
- Abbreviated Early Prolonged Exposure Therapy (Experimental): AEPET, including Manualized Resilience-Based supportive Therapy.
  Interventions: Behavioral: Abbreviated Early Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Abbreviated Early Prolonged Exposure Therapy — Since many trauma patients are discharged within 4 weeks, AEPET with the same length (45 minutes - 1 hour) and number of sessions as PET, is given in a shorter time period (daily for 3 days as opposed to weekly over 3 weeks).
  Arms: Abbreviated Early Prolonged Exposure Therapy

SUMMARY:
The objective of this study is to assess the feasibility and effectiveness of AEPET plus Resilience Based Therapy (RBT) versus RBT alone for the prevention of PTSD and depression in trauma patients. The intervention group who have AEPET plus RBT will have reduced level of post traumatic stress symptoms and depression post sessions as well as reduced symptoms of PTSD and depression at 4- 6 weeks as compared to the control group who have -"Resilience Based" less specific supportive therapy.

DETAILED DESCRIPTION:
Background:

The Sunnybrook Health Sciences Centre contains one of the largest trauma centers in Canada, treating approximately 1,100 patients annually. Many of these cases typically include unexpected events that can cause severe or life-threatening injuries and at the time patients often experience horror and helplessness and even threat of death. Many of these traumatic injuries are not only physically damaging but psychologically as well. Lower psychological well-being has been reported in trauma survivors, specifically symptoms related to Depression and Post Traumatic Stress Disorder (PTSD).

Methods:

Patients in trauma units admitted within the previous week will be approached by a trauma team member to see if they are willing to be approached by a Research Assistant (RA). If they agree, an RA will seek permission to screen for eligibility and complete recruitment and the informed consent process. Patients will be recruited if they have a premorbid risk factor for PTSD or if their current trauma resulted in clear memories of it being life threatening and horrifying to them or resulted in dissociation. Participants will be excluded if they were intoxicated at the time of the trauma, they seem cognitively impaired or if they suffered a severe head injury.

After stratified 1:1 randomization to either AEPET plus RBT (n=10-15) or RBT alone (n=10-15) , consenting participants will complete baseline measures and 3 therapy sessions, starting within 1 week post-trauma. Participants will be scheduled for their first 30-60 minute therapy session at consent . Participants will receive two more face-to-face / telephone sessions as close together as possible, followed by completing three questionnaires after the second session.

In the protocol, participants will give consent within 1 week post-trauma. Eligible participants will be recruited if they are expected to remain in hospital for a minimum of 1 day to be able to complete 1 of the 3 sessions. If a patient is discharged before the second or third / final therapy session, they will be phoned for two or one remaining sessions, respectively.

Participants will be included as 'treated' in the data analysis if they complete 2 out of the 3 therapy treatments.

TAU will include routine psychosocial care, psychological management of trauma patients, including brief assessment and referral to psychiatry if the trauma team thinks it's necessary. RBT will specifically address the five essential intervention principles for the psychosocial management of trauma which include promotion of safety, self-efficacy, calming, connectedness and hope.

The following questionnaires will be administered to patients in both the control and intervention group at baseline,

1. Stanford Acute Stress Reaction Questionnaire (SASRQ)
2. Posttraumatic Cognitions Inventory (PTCI)
3. Beck Depression Inventory II (BDI-II)

The following questionnaires will be administered to patients in both the control and intervention group at baseline, with instructions to complete after their second therapy session:

1. Stanford Acute Stress Reaction Questionnaire (SASRQ)
2. Posttraumatic Cognitions Inventory (PTCI)
3. Beck Depression Inventory II (BDI-II)

The following questionnaire will be administered by phone (1,2) and sent by mail (3, 4) to patients one month post enrollment in the study:

1. (by phone) Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
2. (by phone) PTSD Symptom Scale interview (PSSI)
3. (by mail) Posttraumatic Cognitions Inventory (PTCI)
4. (by mail) Beck Depression Inventory II (BDI-II)

Planned Data Analysis:

Data will be analyzed using SAS. Descriptive statistics will be calculated for all variables. Bivariate comparisons of variables will be made using χ2, Spearman and Pearson correlation coefficients, Student t tests and ANOVA. Stepwise multivariable regression analyses will be undertaken to examine significant correlates of PTSD and between group (control and intervention) differences in all the outcomes. Statistical tests will be two tailed with alpha set at 0.05.

The anticipated outcomes include lower levels of PTSD and depressive symptoms for those having AEPET + RBT vs. RBT alone by self report and by semi structured interview at 4-6 weeks.

Significance:

In testing the feasibility and effectiveness of AEPET as a novel treatment for the prevention of PTSD within its trauma ward, Sunnybrook Hospital would potentially pioneer a feasible and cost-effective method for employing a quicker response, targeted treatment for mitigating symptoms of PTSD and depression after trauma.

ELIGIBILITY:
Inclusion Criteria

1. Age 17-75
2. Experienced an acute physical trauma in the past 4 days where the patient believed it was potentially life-threatening in their mind at the time of the trauma
3. Have some clear memories of the trauma
4. Contain any risk factors for PTSD
5. An abbreviated Injury Severity (AIS) score of 1-3 (Minor, Moderate and Severe; not life threatening)

Exclusion Criteria

1. Inability to communicate sufficiently in English to be able to complete questionnaires and provide informed consent
2. A diagnosis of psychosis, mental retardation or autism
3. Blood alcohol level of >0.08mmol/L (25 mg/dl) at time of admission
4. Cognitive impairment apparent on interview/collateral from trauma team
5. Severe head injury

Withdrawal Criteria

1. If the patient is thought to be at risk to self or others, or be in need of immediate psychiatric assessment, in which case the patient will be referred urgently for assessment with psychosocial oncology or department of psychiatry
2. If the patient wishes to discontinue the study
3. If the patient is noted to be cognitively impaired during the course of the study such that he/she cannot complete a questionnaire reliably or physically impaired such that it is too burdensome for the patient to complete the questionnaire package.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
PTSD Presence and Severity at 1 month follow-up | 1 - 2 Months
  Scale used to assess presence and measure severity: The Post-Traumatic Stress Disorder (PTSD) Symptom Scale -Interview (PSS-I)

SECONDARY OUTCOMES:
Change from Baseline Trauma-related Thoughts and Beliefs at Therapy Time-Point 2 and 1 month follow-up | 1 - 2 Months
  Scale used to measure Trauma-related Thoughts and Beliefs: The Posttraumatic Cognitions Inventory (PTCI)
Change from Baseline Depresssive Symptoms at Therapy Time-Point 2 and 1 month follow-up | 1 - 2 Months
  Scale used to measure Depressive Symptoms: Beck Depression Inventory II (BDI-II)
PTSD Presence and Severity and Diagnosis at 1 month follow-up | 1 - 2 Months
  Scale used to assess presence and measure severity of PTSD: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Psychological Well-being at 1 month follow-up | 1 - 2 Months
  Scale used to measure Psychological Well-being: The Stanford Acute Stress Reaction Questionnaire (SASRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Ellis, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada